CLINICAL TRIAL: NCT07340619
Title: UNLOCK - EPIBREAST, a Phase II Study of Prifetrastat (PF-07248144), a KAT6 Inhibitor, Plus Fulvestrant for Advanced HR+/HER2- Breast Cancer, With Biomarkers Analyses
Brief Title: Clinical Trial Evaluating the Biological Activity of a New Drug Identified as Prifetrastat (PF-07248144), Combined With Fulvestrant for the Treatment of Patients With Hormone Receptor Positive (HR+) and HER2 Negative (HER2-) Breast Cancer Extended to Other Organs.
Acronym: EPIBREAST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UC-GMP-2504; 2025-521982-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Metastatic (Stage IV) Melanoma
Keywords: Epiddrug; breast cancer RH+ /HER2-; KAT6 inhibitor; prifetrastat; PF-07248144
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 : prifetrastat monotherapy for 15days then combination with fulvestrant (Experimental): Patients will receive prifetrastat 5mg QD monotherapy for 2 weeks and then combination of prifetrastat 5mg QD plus fulvestrant 500-mg intramuscular injection on day 15 cycle 1, on day 1 and day 15 of cycle 2 and then on day 15 of subsequent 28-day (±3 days) cycles.
  In both cohorts, men and premenopausal women will receive in addition a LH-RH analogue (goserelin, leuprorelin or triptorelin) every 28 days ±3 days, as per standard practice. Administration schedule of the analogue will follow the same schedule as described for fulvestrant, which depends on the allocated cohort.
  Interventions: Drug: prifetrastat monotherapy for 15 days then combination with fulvestrant
- Cohort 2 : prifetrastat incombination with fulvestrant (Experimental): Patients will receive combination prifetrastat 5mg QD plus fulvestrant 500-mg intramuscular injection on days 1 and 15 of cycle 1 and on day 1 of subsequent 28-day (±3 days) cycles.
  In both cohorts, men and premenopausal women will receive in addition a LH-RH analogue (goserelin, leuprorelin or triptorelin) every 28 days ±3 days, as per standard practice. Administration schedule of the analogue will follow the same schedule as described for fulvestrant, which depends on the allocated cohort.
  Interventions: Drug: prifetrastat in combination with fulvestrant

INTERVENTIONS:
Drug: prifetrastat monotherapy for 15 days then combination with fulvestrant — Patients will receive prifetrastat 5mg QD monotherapy for 2 weeks and then combination of prifetrastat 5mg QD plus fulvestrant 500-mg intramuscular injection on day 15 cycle 1, on day 1 and day 15 of cycle 2 and then on day 15 of subsequent 28-day (±3 days) cycles.
  Arms: Cohort 1 : prifetrastat monotherapy for 15days then combination with fulvestrant
Drug: prifetrastat in combination with fulvestrant — Patients will receive combination prifetrastat 5mg QD plus fulvestrant 500-mg intramuscular injection on days 1 and 15 of cycle 1 and on day 1 of subsequent 28-day (±3 days) cycles
  Arms: Cohort 2 : prifetrastat incombination with fulvestrant

SUMMARY:
Although treatments for breast cancer have improved, 20-30% of patients with early disease develop metastases (cancer that spreads to other parts of the body). Among the different types of breast cancer, hormone-sensitive cancers that do not overexpress the HER2 protein (HR+/HER2-) are the most common. For patients with this type of cancer, an endocrine treatment such as aromatase inhibitors, tamoxifen or fulvestrant, is often used and may be combined with drugs called CDK4/6 inhibitors, which help improve survival rate. However, when the cancer becomes resistant to these treatments, treatment strategies are more limited

A new drug, prifetrastat (PF-07248144), which targets KAT6 proteins, which play a role in the growth of cancer cells, has shown promising results. Indeed, associated with fulvestrant, it allowed to fight against cancer in some patients who had already received many treatments.

The UNLOCK-EPIBREAST study aims to investigate whether the combination of prifetrastat plus fulvestrant could offer a new therapeutic option for people with HR+/HER2- metastatic breast cancer who have already received endocrine therapy plus CDK4/6 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the trial, all patients must meet all the following criteria:

1. Patient must have signed the written informed consent prior to any study specific screening procedures.

   Note : When the patient is physically unable to give her/his written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Adult participants age ≥18 years.
3. Histological or cytological diagnosis of advanced or metastatic ER+HER2- breast cancer.
4. Participants must have progressive disease after at least 1 prior line of a CDK4/6 inhibitor and at least 1 prior line of endocrine therapy received in metastatic setting. Participants must not have received more than 3 prior lines of systemic therapies including up to 2 lines of cytotoxic chemotherapy for visceral disease in advanced or metastatic setting. Note that prior treatment with fulvestrant is permitted.
5. Participants must have documentation of ER-positive tumor (≥10% positive stained cells) based on most recent tumor biopsy utilizing an assay consistent with local standards.
6. Participants must have documentation of HER2-negative tumor: HER2-negative tumor is determined as immunohistochemistry score 0/1+ or HER2 2+ and negative by in situ hybridization (FISH/CISH/SISH/DISH) defined as a HER2/CEP17 ratio <2 or for single probe assessment a HER2 copy number <4.
7. Female participants with premenopausal status (see section 5.8.4) must be willing to undergo medically induced menopause by treatment with approved LHRH agonist such as goserelin, leuprolide or equivalent agents to induce chemical menopause.
8. Participants must have at least 1 measurable lesion as defined by RECIST version 1.1 that has not been previously irradiated.
9. Participants must present with a metastatic site easily accessible to a biopsy procedure and be a non-bone and non-irradiated site.
10. ECOG Performance Status PS 0 or 1.
11. Expected survival of more than 3 months.
12. Adequate bone marrow function, including:

    1. ANC ≥1,500/mm3 or ≥1.5 x 109/L;
    2. Platelets ≥100,000/mm3 or ≥100 x 109/L;
    3. Hemoglobin ≥9 g/dL.
13. Adequate renal function, including serum creatinine ≤1.5 x ULN or estimated creatinine clearance GFR ≥50 mL/min as calculated using the method standard for the institution. In equivocal cases, a 24-hour urine collection test can be used to estimate creatinine clearance more accurately.
14. Adequate liver function, including:

    1. Total serum bilirubin ≤1.5 x ULN unless the participant has documented Gilbert syndrome;
    2. AST and ALT ≤2.5 x ULN; AST and ALT ≤5.0 x ULN if there is liver involvement.
15. Adequate blood clotting function: International Normalized Ratio (INR)/Prothrombin Time (PT) and either partial thromboplastin Time (PTT) or activated Partial Thromboplastin Time (aPTT) ≤1.5 x ULN.
16. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1 except for AEs not constituting a safety risk by investigator judgment.
17. Participants must consent to the use of their archived and/or collected tumor specimen, as well as blood samples, as detailed in the protocol, for future scientific research which includes, but is not limited to DNA, RNA, and protein-based biomarker detection.
18. Women of childbearing potential must have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) result within 3 days of enrolment.
19. Men or women of childbearing potential must agree to the use of effective contraceptive for the study duration and for at least 28 days after the last dose of study treatment for women, and at least 93 days for men.
20. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
21. . Patients must be affiliated to a Social Security System (or equivalent).
22. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion criteria:

Patients are not eligible to participate if they meet any of the following criteria:

1. Participants with known symptomatic brain metastases requiring steroids. Participants with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to randomization, have discontinued corticosteroid treatment for these metastases for at least 3 weeks and are neurologically stable for 2 months (requires MRI confirmation).
2. Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term (including participants with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement). Note: Participants with indwelling catheter for drainage, or requirement for drainage no more frequently than once a month will be allowed.
3. Participants with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ. Other indolent cancers that do not interfere with assessment of primary cancer under study may be allowed with prior sponsor approval.
4. Major surgery within 3 weeks prior to randomization.
5. Radiation therapy within 3 weeks prior to randomization.
6. Systemic anti-cancer therapy within 3 weeks prior to randomization. If the last immediate anti-cancer treatment contained an antibody-based agent(s) (approved or investigational), then an interval of 28 days or 5 half-lives (whichever is shorter) of the agent(s) prior to receive the study intervention treatment is required.
7. Prior irradiation to >25% of the bone marrow.
8. Participants with active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) HBV, HCV, known HIV or AIDS related illness. HIV seropositive subjects who are healthy and low risk for AIDS-related outcomes could be considered eligible.

   Eligibility criteria for HIV-positive subjects should be evaluated and discussed with sponsor's medical monitor and will be based on current and past CD4 and T-cell counts, history (if any) of AIDS-defining conditions (eg, opportunistic infections), and status of HIV treatment. Also, the potential for drug-drug interactions will be taken into consideration. In equivocal cases, with positive serology, those participants with a negative viral load are potentially eligible provided the other entry criteria are met.
9. Unmanageable ascites (limited medical treatment to control ascites is permitted, but all participants with ascites require review by sponsor's medical monitor).
10. Baseline 12 -lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >470 msec, complete LBBB, signs of an acute myocardial infarction, ST changes suggestive of active myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >470 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF- should be used for decision making and reporting. If QTcF exceeds 470 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer -interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants. Cases must be discussed in detail with sponsor's medical monitor to judge eligibility.
11. Any of the following in the previous 6 months: myocardial infarction, long QT syndrome, Torsade de Pointes, clinically important atrial or ventricular arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), serious conduction system abnormalities (eg, bifascicular block [defined as right bundle branch and left anterior or posterior hemiblock], 3rd degree AV block), unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF, New York Heart Association class III or IV, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, and/or other clinical significant episode of thrombo embolic disease and ongoing cardiac dysrhythmias of NCI CTCAE ≥Grade 2. For Grade 2 atrial fibrillation, may be considered eligible with sponsor approval (e.g if improved to Grade 1 with non-urgent medical intervention or chronic Grade 2 atrial fibrillation with good rate control with non-urgent medical intervention). If a participant has a cardiac rhythm device/pacemaker placed and QTcF >470 msec, the participant can be considered eligible. Participants with cardiac rhythm device/pacemaker must be discussed in detail with sponsor's medical monitor to judge eligibility.
12. Therapeutic anticoagulation.
13. Hypertension that cannot be controlled by optimal medical therapy (eg, ≥160/100 mmHg).
14. Participation in other studies involving investigational drug(s) within 3 weeks prior to study entry. Participation in observational or in long term follow-up of other studies is allowed if no procedures which may interfere with the interpretation of study results will be performed.
15. Known or suspected hypersensitivity or severe allergy to active ingredient/excipients of study drug(s) such as lactose.
16. Prior treatment with prifetrastat. Note that prior treatment with fulvestrant is permitted.
17. Active inflammatory GI disease, refractory and unresolved chronic diarrhea or previous gastric resection, lap band surgery or other GI conditions and surgeries that may significantly alter the absorption of prifetrastat. Gastroesophageal reflux disease under treatment is allowed.
18. Current use or anticipated need for food or drugs that are known moderate or strong CYP3A4/5 inhibitors, including their administration within 10 days or 5 half-lives of the CYP3A4/5 inhibitor, whichever is longer prior to first dose of study intervention (see Appendix 8 for a list of exemplary strong/moderate CYP3A4/5 inhibitors).
19. Current use or anticipated need for food or drugs that are known strong CYP3A4/5 inducers, including their administration within 10 days or 5 half-lives of the CYP3A4/5 inducer, whichever is longer prior to the first dose of study intervention (see Appendix 8 for a list of exemplary strong/moderate CYP3A4/5 inducers).
20. Current use or anticipated need for food or drugs that are known moderate/strong CYP2C9 inhibitors, including their administration within [10 days or 5 half-lives of the CYP2C9 inhibitor, whichever is longer] prior to first dose of investigational product (amiodarone, fluconazole, miconazole, oxandrolone) (see Appendix 8 for a list of exemplary strong/moderate CYP2C9 inhibitors).
21. Current use or anticipated need for drugs that are known moderate/strong CYP2C9 inducers, including their administration within [10 days or 5 half-lives of the CYP2C9 inducer, whichever is longer] prior to the first dose of investigational product (carbamazepine, rifampin) (see Appendix 8 for a list of exemplary strong/moderate CY2C9 inducers).
22. Patient is currently pregnant, breastfeeding, or planning to become pregnant.
23. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
24. Patient unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
25. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male, female
Enrollment: 51 (Estimated)
Dates: Start 2026-05-18 (Estimated); Primary Completion 2028-11-18 (Estimated); Study Completion 2029-11-18 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the effect of prifetrastat with fulvestrant on ctDNA-based mutation burden among patients with HR+/HER2- mBC. | From first treatment administration to disease progression or death, up to 5 years
  A Guardant Health (Guardant360® CDx) assay will be used for ctDNA detection and sequencing and evaluation of tumor mutation burden defined by the mean change in Variant Allele Frequency (VAF) of 74 prespecified genes, from cycle 1 to cycle 3.
  Primary endpoint will be evaluated per cohort (as defined in section "Therapeutic regimen" below) and in the overall population.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin VERRET, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Fabrice ANDRE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris

IPD SHARING:
Plan to Share IPD: No